CLINICAL TRIAL: NCT03007355
Title: The Use of Peripheral Perfusion Index as a Predictor for Patient's Response to Deliberate Hypotension During Functional Endoscopic Sinus Surgery A Prospective Observational Study
Brief Title: Peripheral Perfusion Index (PPI) as Monitor During Deliberate Hypotensive Anesthesia
Acronym: PPI
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Abeer Ahmed, MD, Lecturer of Anesthesia - Faculty of Medicine, Cairo University
Other Study IDs: N 2015
Record Dates: First submitted 2016-12-26; First posted 2017-01-02 (Estimated); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Monitoring During Deliberate Hypotensive Anesthesia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: peripheral perfusion index measurement

SUMMARY:
Hypotensive anesthesia is effective in reducing the intraoperative blood loss. The risk of hypoperfusion of vital organs continues to be a concern. An adequate monitoring of tissue perfusion and oxygenation is crucial issue. Peripheral Perfusion Index (PPI) as a noninvasive new monitoring, can reflect the peripheral perfusion dynamics.

This study is designed to explore the behaviour and trend of PPI during nitroglycerine induced deliberate hypotensive anesthesia in adult patients undergoing functional endoscopic sinus surgery (FESS).

ELIGIBILITY:
Inclusion Criteria:

* Patients, aged from 18-50 years, ASA physical status I and II, undergoing functional endoscopic sinus surgery (FESS) under deliberate hypotensive anesthesia

Exclusion Criteria:

* Patients with systemic hypertension, cardiovascular disease, cerebrovascular insufficiency, coagulation defects, renal or hepatic insufficiency, and hypersensitivity to the study drugs will be excluded from the study. Patients receiving vasoactive drugs or beta blockers will be also excluded from the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: adult male or females, aged between 18-50 years, ASA class I ans II
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2017-01; Primary Completion 2017-10 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
correlation between PPI and T1 | start of nitroglyceirn infusion till target arterial pressure is reached up to 2 hours
  correlation of baseline values of PPI and time required to achieve target mean arterial pressure.